CLINICAL TRIAL: NCT02223676
Title: Is Length of Stay in the Emergency Department Reduced When Clinical Pharmacists Conduct Medication History? - a Cluster Randomized Study
Brief Title: Clinical Pharmacists in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Randers Regional Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1-16-02-379-13
Record Dates: First submitted 2014-01-07; First posted 2014-08-22 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2014-08

CONDITIONS: Medication Reconciliation
Keywords: Pharmacy; Length-of-stay; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Clinical pharmacists conduct medication history
  Interventions: Procedure: Clinical pharmacists conduct medication history
- Control (No Intervention): standard procedures for admission is followed

INTERVENTIONS:
Procedure: Clinical pharmacists conduct medication history — pharmacists conduct medication history before the physician interviews the patient and does not spend time on conducting medical history
  Arms: Intervention

SUMMARY:
The purpose of this study is to investigate the effect of implementing clinical pharmacists in the Emergency Department Team at Randers Regional Hospital. The clinical pharmacists conduct medication history, make medical interaction screenings, -reconciliations and -reviews on unscheduled patients admitted to the Emergency Department during daytime.

ELIGIBILITY:
Inclusion Criteria:

* unscheduled patients admitted to the Emergency Department at Randers Regional Hospital at weekdays during daytime (9 am to 16.15 pm)
* 4 or more drugs prescribed

Exclusion Criteria:

* patients triage red
* patients who cannot give informed consent
* terminal patients
* patients admitted to detoxification
* patients refered to the acute outpatient department
* patients remaining in the Emergency Department overnight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Emergency Department Length of stay | From arrival to the Emergency Department to either admission or discharge, which in average will be 6 hours.

SECONDARY OUTCOMES:
Time from patient arrival to the treatment schedule is ready | From arrival to the Emergency Department to either admission or discharge, which in average will be 6 hours.
Patient safety | From arrival to the Emergency Department to either admission or discharge, which in average will be 6 hours.
  Number of recommended changes in drugs or dosage per patient. The changes are rated according to a PCNE-classification for drug-related problems.

OTHER OUTCOMES:
The impact of the intervention in the Emergency Department on the existing medication review by clinical pharmacist at the acute ward | 1-3 days after admission to Emergency Department when the secondary medication review takes place
  We estimate whether the intervention is time-saving (by recording and comparing time spent for secondary/excisting medication review at the acute ward between patients allocated to the intervention and control group, respectively) and reduce the workload of the clinicians (number and kind of interventions at secondary medication review in the two groups)
The impact of the intervention in the Emergency Department on the dispensing of medicine (done by nurses) | During actual admission to the Emergency Department and the period after inclusion of patients
  time used and the possibility of substitutions

CONTACTS AND LOCATIONS:
Locations (1):
- Randers Regional Hospital, Randers, Region Midt, Denmark